CLINICAL TRIAL: NCT06069466
Title: Epidemiological Characteristics and Prediction System of Acute Respiratory Distress Syndrome in China RICUs-CHARDS II Study
Brief Title: Epidemiological Characteristics and Prediction System of Acute Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Huang Xu, associate chief physician, China-Japan Friendship Hospital
Other Study IDs: 2023-NHLHCRF-YYPP-TS-04
Record Dates: First submitted 2023-10-02; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; mortality; incidence; prognosis; predictive model; AI
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Transcriptome mRNA of blood and BALF
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS patient

SUMMARY:
This project intends to adopt the multicenter prospective real-world study method to conduct a preliminary study on the incidence, grading, risk factors, respiratory support strategies, in-hospital mortality, 3-month mortality, 6-month mortality, 1-year mortality, quality of life, lung function and limb function recovery, cognitive function, return to work and other conditions of ARDS patients in RICU. By collecting 1,000 patients, a clinical database related to ARDS in China was established to provide essential data and ideas for promoting standardized diagnosis and treatment technology for ARDS patients and further clinical intervention research. At the same time, ARDS biobank was established in China-Japan Hospital and Xiangya Hospital to realize the integration of clinical data and sample resources, and the prediction model of ARDS survival and complications of tuberculosis clinical data and biological samples was established by using big data and AI technology.

ELIGIBILITY:
Inclusion Criteria:

* New or worsening respiratory symptoms less than 7 days after the acute blow.
* CT/X-ray: Double lung infiltration that cannot be fully explained by pleural effusion, lobar/whole atelectasis, and nodule.
* Respiratory failure that cannot be explained by heart failure or fluid overload
* After 15min assisted ventilation (PEEP or CPAP ≥ 5cmH2O) or HFNC with flow≥30L/min, PaO2/FiO2≤300mmHg
* Classification of ARDS: mild (200mmHg < PaO2/FIO2 ≤ 300mmHg), moderate (100mmHg < PaO2/FIO2 ≤ 200mmHg), and severe (PaO2/FIO2 ≤ 100mmHg) and 4 ancillary variables for severe ARDS

Exclusion Criteria:

* younger than 18 years old
* Patients or family members refused to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with ARDS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
the prognosis of ARDS patients | from 28d to 1 year
  ICU mortality, 28-day mortality, 90-day mortality and 1-year mortality of ARDS patients

SECONDARY OUTCOMES:
Incidence of ARDS in ICUs | 2 years
  Incidence of ARDS in ICUs
Length of hospital stay in ARDS patients | during hospitalization
  Length of hospital stay in ARDS patients
VFDs within 28 days | 28 days
  Mechanical ventilation free days within 28 days
Long-term quality of life and long-term lung function | 1 year
  3month，6month，1year quality of life score and 1year lung function
Rates of mechanical ventilation strategies are consistent with guidelines rates of rates of mechanical ventilation strategies consistent with guidelines | during hospitalization
  consistence of lung protective ventilation strategies（including small tidal volume and limitation of Pplat）
Survival risk factors in hospitalized ARDS patients | during hospitalization
  Survival risk factors in hospitalized ARDS patients
Risk factors for ARDS complications | during hospitalization
  Risk factors for ARDS complications（including AKI and barotrauma）

CONTACTS AND LOCATIONS:
Overall Officials: Xu Huang, PhD, Principal Investigator — Department of Respiratory and Critical Care Medicine, China-Japan Friendship Hospital
Locations (1):
- Department of Pulmonary and Critical Care Medicine, Center of Respiratory Medicine, China-Japan Friendship Hospital, Beijing, Beijing Municipality, China